CLINICAL TRIAL: NCT02547649
Title: A Multicenter, Double-Blind Study of the Safety, Tolerability, and Immunogenicity of V114 Compared to Prevnar 13™ in Healthy Pneumococcal Vaccine-Naïve Adults 50 Years of Age or Older
Brief Title: Safety, Tolerability, and Immunogenicity of Two Formulations of V114 in Healthy Adults 50 Years of Age or Older (V114-006)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V114-006; V114-006 (Other: Merck Protocol Number)
Record Dates: First submitted 2015-09-10; First posted 2015-09-11 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- V114 Formulation A (Experimental): Participants receive a single 0.5 mL intramuscular injection of V114 Formulation A on Day 1
  Interventions: Biological: V114-A
- V114 Formulation B (Experimental): Participants receive a single 0.5 mL intramuscular injection of V114 Formulation B on Day 1
  Interventions: Biological: V114-B
- Prevnar 13® (Active Comparator): Participants receive a single 0.5 mL intramuscular injection of Prevnar 13® on Day 1
  Interventions: Biological: Prevnar 13®

INTERVENTIONS:
Biological: V114-A — Formulation A of V114 contains 2 µg of pneumococcal capsular polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19F, 19A, 22F, 23F, and 33F; 4 µg of serotype 6B; 32 µg of CRM197 protein carrier; and 125 µg of Aluminum Phosphate Adjuvant in each 0.5 mL dose (V114-A uses a unique excipient to improve stability of the vaccine against physical stress).
  Arms: V114 Formulation A
Biological: V114-B — Formulation B of V114 contains 2 µg of pneumococcal capsular polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19F, 19A, 22F, 23F, and 33F; 4 µg of serotype 6B; 32 µg of CRM197 protein carrier; and 125 µg of Aluminum Phosphate Adjuvant in each 0.5 mL dose (V114-B uses a unique excipient to improve stability of the vaccine against physical stress).
  Arms: V114 Formulation B
Biological: Prevnar 13® — Pneumococcal capsular polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 23F (2.2 mcg each), and 6B (4.4 mcg) in each 0.5 mL dose.
  Arms: Prevnar 13®

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and immunogenicity of a single dose of different formulations of V114 (V114-A and V114-B) and Prevnar 13® (pneumococcal 13-valent conjugate vaccine) in adult participants

≥50 years of age in good health.

ELIGIBILITY:
Inclusion Criteria:

* Good health; any underlying chronic illness must be documented to be in stable condition
* Highly unlikely to conceive through 6 weeks after administration of the study vaccine

Exclusion Criteria:

* Prior administration of any pneumococcal vaccine
* History of invasive pneumococcal disease (IPD) [positive blood culture, positive cerebrospinal fluid culture, or other sterile site) or known history of other culture-positive pneumococcal disease
* Known hypersensitivity to any vaccine component
* Known or suspected impairment of immune function
* Received systemic corticosteroids for >=14 consecutive days and has not completed treatment <=30 days prior to study entry, or received systemic corticosteroids exceeding physiologic replacement doses within 14 days prior to study vaccination
* Coagulation disorder contraindicating intramuscular vaccination
* Receives immunosuppressive therapy, including chemotherapeutic agents used to treat cancer or other conditions, and treatments associated with organ or bone marrow transplantation, or autoimmune disease
* Received a blood transfusion or blood products, including immunoglobulins within the 6 months before receipt of study vaccine or is scheduled to receive a blood transfusion or blood product within 30 days of receipt of study vaccine. Autologous blood transfusions are not considered an exclusion criterion.
* Participated in another clinical study of an investigational product within 2 months before the beginning of or any time during the duration of the current clinical study
* Breast feeding
* User of recreational or illicit drugs or has had a recent history (within the last year) of drug or alcohol abuse or dependence

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 690 (Actual)
Dates: Start 2015-10-08 (Actual); Primary Completion 2016-01-20 (Actual); Study Completion 2016-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Stacey HL, Rosen J, Peterson JT, Williams-Diaz A, Gakhar V, Sterling TM, Acosta CJ, Nolan KM, Li J, Pedley A, Benner P, Abeygunawardana C, Kosinski M, Smith WJ, Pujar H, Musey LK. Safety and immunogenicity of 15-valent pneumococcal conjugate vaccine (PCV-15) compared to PCV-13 in healthy older adults. Hum Vaccin Immunother. 2019;15(3):530-539. doi: 10.1080/21645515.2018.1532249. Epub 2019 Jan 16. PMID 30648919

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy, pneumococcal vaccine-naïve adults ≥50 years of age were recruited at 23 sites in the United States.
Groups:
- V114-A: Participants receive a single 0.5 mL intramuscular injection of V114 Formulation A on Day 1. Formulation A of V114 contains 2 µg of pneumococcal capsular polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19F, 19A, 22F, 23F, and 33F; 4 µg of serotype 6B; 32 µg of CRM197 protein carrier; and 125 µg of Aluminum Phosphate Adjuvant in each 0.5 mL dose (V114-A uses a unique excipient to improve stability of the vaccine against physical stress).
- V114-B: Participants receive a single 0.5 mL intramuscular injection of V114 Formulation B on Day 1. Formulation B of V114 contains 2 µg of pneumococcal capsular polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19F, 19A, 22F, 23F, and 33F; 4 µg of serotype 6B; 32 µg of CRM197 protein carrier; and 125 µg of Aluminum Phosphate Adjuvant in each 0.5 mL dose (V114-B uses a unique excipient to improve stability of the vaccine against physical stress).
- Prevnar 13®: Participants receive a single 0.5 mL intramuscular injection of Prevnar 13™ on Day 1.
Period: Overall Study
Arm/Group | V114-A | V114-B | Prevnar 13®
Started (Randomized) | 231 | 231 | 228
Vaccinated | 231 | 231 | 227
Completed | 228 | 226 | 224
Not Completed | 3 | 5 | 4
Not completed — Lost to Follow-up | 3 | 1 | 1
Not completed — Not vaccinated | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 4 | 2

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population consists of all vaccinated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | V114-A | V114-B | Prevnar 13® | Total
Number analyzed (Participants) | 231 | 231 | 227 | 689
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.4 (8.3) | 63.4 (8.3) | 63.1 (8.1) | 63.3 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 126 | 133 | 385
  Male | 105 | 105 | 94 | 304

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Adverse Event (AE)
Description: The percentage of participants experiencing ≥1 AE(s) in each arm was determined. An AE is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 14 days after vaccination
Population: All participants who received study vaccination are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114-A | V114-B | Prevnar 13®
Number analyzed (Participants) | 231 | 231 | 227
Percentage of Participants | 74.9 | 72.3 | 67.4

2. Primary Outcome: Percentage of Participants With a Solicited Injection-site Adverse Event (AE)
Description: The percentage of participants experiencing ≥1 solicited injection-site AE(s) in each arm was determined.
Time Frame: Up to 14 days after vaccination
Population: All participants who received study vaccination are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114-A | V114-B | Prevnar 13®
Number analyzed (Participants) | 231 | 231 | 227
Percentage of Participants
  Erythema | 8.7 | 11.3 | 10.1
  Pain | 62.3 | 60.2 | 52.4
  Swelling | 11.7 | 16.5 | 12.3

3. Primary Outcome: Percentage of Participants With a Solicited Systemic Adverse Event (AE)
Description: The percentage of participants experiencing ≥1 solicited systemic AE(s) in each arm was determined.
Time Frame: Up to 14 days after vaccination
Population: All participants who received study vaccination are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114-A | V114-B | Prevnar 13®
Number analyzed (Participants) | 231 | 231 | 227
Percentage of Participants
  Arthralgia | 9.5 | 7.4 | 6.2
  Myalgia | 22.9 | 18.6 | 14.1
  Headache | 12.1 | 12.6 | 16.7
  Fatigue | 24.2 | 17.7 | 22.5

4. Primary Outcome: Percentage of Participants With a Serious Adverse Event (SAE)
Description: The percentage of participants experiencing ≥1 SAE(s) in each arm was determined.
Time Frame: Up to 30 days after vaccination
Population: All participants who received study vaccination are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114-A | V114-B | Prevnar 13®
Number analyzed (Participants) | 231 | 231 | 227
Percentage of Participants | 0.4 | 0.9 | 0.0

5. Primary Outcome: Percentage of Participants With Vaccine-Related Serious Adverse Event (SAE)
Description: The percentage of participants experiencing ≥1 vaccine-related SAEs(s) in each arm was determined.
Time Frame: Up to 30 days after vaccination
Population: All participants who received study vaccination are included.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114-A | V114-B | Prevnar 13®
Number analyzed (Participants) | 231 | 231 | 227
Percentage of Participants | 0.0 | 0.0 | 0.0

6. Primary Outcome: Geometric Mean Titers (GMTs) of Serotype-specific Opsonophagocytic Killing Activity (OPA) at One Month Post-Vaccination
Description: The OPA GMTs of each common serotype (CS) and V114-specific serotype (VS) were determined in each arm. Titer levels were determined with the multiplexed opsonophagocytic assay (MOPA).
Time Frame: Day 30 (one month after vaccination)
Population: All vaccinated participants with data available are included.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | V114-A | V114-B | Prevnar 13®
Number analyzed (Participants) | 231 | 231 | 227
Titers
  CS1: number analyzed (Participants) | 209 | 203 | 204
  CS1 | 196.79 [145.49 to 266.17] | 144.01 [106.06 to 195.54] | 127.19 [93.19 to 173.60]
  CS3: number analyzed (Participants) | 206 | 203 | 199
  CS3 | 104.78 [83.69 to 131.18] | 61.41 [48.99 to 76.97] | 33.10 [25.41 to 43.12]
  CS4: number analyzed (Participants) | 213 | 206 | 210
  CS4 | 1314.31 [1050.53 to 1644.31] | 929.53 [722.68 to 1195.57] | 1195.73 [931.75 to 1534.49]
  CS5: number analyzed (Participants) | 212 | 204 | 206
  CS5 | 273.79 [201.52 to 372.00] | 269.14 [197.57 to 366.63] | 283.83 [209.93 to 383.74]
  CS6A: number analyzed (Participants) | 214 | 213 | 212
  CS6A | 3849.02 [2937.54 to 5043.31] | 4690.40 [3688.20 to 5964.93] | 4932.72 [3771.98 to 6450.62]
  CS6B: number analyzed (Participants) | 212 | 212 | 208
  CS6B | 4552.54 [3680.12 to 5631.79] | 5082.56 [3984.20 to 6483.72] | 3909.05 [3005.43 to 5084.36]
  CS7F: number analyzed (Participants) | 212 | 210 | 210
  CS7F | 2672.91 [2213.60 to 3227.51] | 2845.64 [2374.74 to 3409.92] | 3659.86 [3036.53 to 4411.14]
  CS9V: number analyzed (Participants) | 215 | 211 | 208
  CS9V | 2514.21 [2014.06 to 3138.57] | 1962.09 [1558.28 to 2470.55] | 2112.91 [1685.97 to 2647.96]
  CS14: number analyzed (Participants) | 214 | 210 | 212
  CS14 | 3496.71 [2776.80 to 4403.25] | 2664.63 [2206.92 to 3217.26] | 3111.50 [2560.29 to 3781.38]
  CS18C: number analyzed (Participants) | 214 | 213 | 209
  CS18C | 1896.14 [1540.37 to 2334.08] | 2687.10 [2169.85 to 3327.65] | 1528.79 [1208.83 to 1933.45]
  CS19A: number analyzed (Participants) | 211 | 213 | 212
  CS19A | 1910.75 [1587.43 to 2299.92] | 2477.75 [2043.94 to 3003.63] | 2045.57 [1692.29 to 2472.59]
  CS19F: number analyzed (Participants) | 210 | 213 | 209
  CS19F | 799.86 [636.72 to 1004.80] | 1084.99 [855.50 to 1376.04] | 810.05 [640.41 to 1024.61]
  CS23F: number analyzed (Participants) | 213 | 206 | 211
  CS23F | 1233.60 [943.88 to 1612.25] | 2198.15 [1702.57 to 2837.99] | 1561.04 [1171.58 to 2079.96]
  VS22F: number analyzed (Participants) | 206 | 204 | 189
  VS22F | 4743.78 [3737.99 to 6020.21] | 3976.66 [3141.02 to 5034.61] | 68.47 [48.39 to 96.88]
  VS33F: number analyzed (Participants) | 212 | 207 | 194
  VS33F | 12457.52 [10076.61 to 15401.00] | 12614.22 [10236.84 to 15543.72] | 2111.66 [1681.43 to 2651.97]

7. Secondary Outcome: Geometric Mean Concentrations (GMCs) of Serotype-specific Immunoglobulin G (IgG) at One Month Post-Vaccination
Description: The IgG GMCs of each common pneumococcal serotype (CS) and V114-specific pneumococcal serotype (VS) were determined for each arm. Concentrations were determined with pneumococcal electrochemiluminescence (PnECL).
Time Frame: Day 30 (one month after vaccination)
Population: All vaccinated participants with data available are included.
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | V114-A | V114-B | Prevnar 13®
Number analyzed (Participants) | 231 | 231 | 227
µg/mL
  CS1: number analyzed (Participants) | 216 | 215 | 214
  CS1 | 5.04 [4.10 to 6.19] | 4.00 [3.34 to 4.79] | 4.15 [3.40 to 5.07]
  CS3: number analyzed (Participants) | 216 | 215 | 214
  CS3 | 0.94 [0.78 to 1.12] | 0.61 [0.51 to 0.72] | 0.48 [0.39 to 0.58]
  CS4: number analyzed (Participants) | 216 | 215 | 214
  CS4 | 1.30 [1.07 to 1.58] | 0.96 [0.79 to 1.16] | 1.39 [1.12 to 1.73]
  CS5: number analyzed (Participants) | 216 | 215 | 214
  CS5 | 3.93 [3.08 to 5.02] | 3.40 [2.66 to 4.34] | 3.37 [2.66 to 4.28]
  CS6A: number analyzed (Participants) | 216 | 215 | 214
  CS6A | 3.88 [2.98 to 5.06] | 4.56 [3.49 to 5.96] | 4.40 [3.29 to 5.88]
  CS6B: number analyzed (Participants) | 216 | 215 | 214
  CS6B | 3.58 [2.78 to 4.63] | 4.71 [3.58 to 6.20] | 3.63 [2.72 to 4.85]
  CS7F: number analyzed (Participants) | 216 | 215 | 214
  CS7F | 4.19 [3.41 to 5.15] | 4.43 [3.59 to 5.47] | 4.69 [3.78 to 5.84]
  CS9V: number analyzed (Participants) | 216 | 215 | 214
  CS9V | 4.17 [3.39 to 5.12] | 3.73 [3.04 to 4.56] | 3.40 [2.74 to 4.22]
  CS14: number analyzed (Participants) | 216 | 215 | 214
  CS14 | 10.54 [8.36 to 13.30] | 6.51 [5.23 to 8.11] | 7.31 [5.79 to 9.22]
  CS18C: number analyzed (Participants) | 216 | 215 | 214
  CS18C | 6.45 [5.21 to 7.98] | 6.51 [5.23 to 8.11] | 7.31 [5.79 to 9.22]
  CS19A: number analyzed (Participants) | 216 | 215 | 214
  CS19A | 8.12 [6.63 to 9.94] | 14.89 [12.20 to 18.18] | 10.42 [8.66 to 12.52]
  CS19F: number analyzed (Participants) | 216 | 215 | 214
  CS19F | 3.96 [3.14 to 4.98] | 7.17 [5.67 to 9.05] | 4.65 [3.81 to 5.68]
  CS23F: number analyzed (Participants) | 216 | 215 | 216
  CS23F | 3.88 [3.03 to 4.97] | 5.49 [4.25 to 7.09] | 4.27 [3.27 to 5.57]
  VS22F: number analyzed (Participants) | 216 | 215 | 214
  VS22F | 3.05 [2.48 to 3.75] | 2.75 [2.25 to 3.36] | 0.25 [0.20 to 0.30]
  VS33F: number analyzed (Participants) | 216 | 215 | 214
  VS33F | 10.28 [8.33 to 12.67] | 7.46 [6.01 to 9.26] | 0.76 [0.60 to 0.96]

8. Secondary Outcome: Percentage of Participants With a ≥4-fold Rise From Baseline in Serotype-specific Opsonophagocytic Killing Activity (OPA) Geometric Mean Titers (GMTs)
Description: The percentage of participants with ≥4-fold rise from baseline in OPA GMTs of each common serotype (CS) and V114-specific serotype (VS) were compared in the V114 and Prevnar® 13 arms. Estimated GMT, GMT ratio, 95% CI, and p-values were obtained from a constrained longitudinal data analysis (cLDA) model.
Time Frame: Baseline and Day 30 (one month after vaccination)
Population: All vaccinated participants with data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114-A | V114-B | Prevnar 13®
Number analyzed (Participants) | 231 | 231 | 227
Percentage of Participants
  CS1: number analyzed (Participants) | 203 | 199 | 201
  CS1 | 70.9 [64.17 to 77.08] | 66.3 [59.31 to 72.86] | 61.7 [54.59 to 68.44]
  CS3: number analyzed (Participants) | 202 | 201 | 195
  CS3 | 71.8 [65.04 to 77.87] | 64.2 [57.13 to 70.80] | 44.1 [37.01 to 51.37]
  CS4: number analyzed (Participants) | 191 | 180 | 185
  CS4 | 84.8 [78.93 to 89.59] | 78.9 [72.19 to 84.61] | 81.6 [75.28 to 86.92]
  CS5: number analyzed (Participants) | 195 | 194 | 198
  CS5 | 68.2 [61.17 to 74.67] | 70.6 [63.67 to 76.93] | 67.2 [60.16 to 73.66]
  CS6A: number analyzed (Participants) | 201 | 199 | 199
  CS6A | 85.1 [79.38 to 89.70] | 82.9 [76.95 to 87.87] | 82.9 [76.95 to 87.87]
  CS6B: number analyzed (Participants) | 185 | 181 | 183
  CS6B | 87.0 [81.31 to 91.51] | 87.3 [81.55 to 91.77] | 84.2 [78.04 to 89.12]
  CS7F: number analyzed (Participants) | 187 | 191 | 188
  CS7F | 67.9 [60.71 to 74.54] | 74.3 [67.54 to 80.38] | 75.0 [68.18 to 81.02]
  CS9V: number analyzed (Participants) | 195 | 188 | 190
  CS9V | 64.6 [57.46 to 71.31] | 59.6 [52.19 to 66.65] | 60.5 [53.19 to 67.53]
  CS14: number analyzed (Participants) | 198 | 197 | 205
  CS14 | 61.6 [54.46 to 68.42] | 50.3 [43.06 to 57.44] | 48.3 [41.28 to 55.36]
  CS18C: number analyzed (Participants) | 191 | 185 | 185
  CS18C | 74.9 [68.10 to 80.85] | 73.0 [65.97 to 79.23] | 64.3 [56.96 to 71.22]
  CS19A: number analyzed (Participants) | 187 | 196 | 197
  CS19A | 74.9 [68.02 to 80.91] | 73.0 [66.17 to 79.04] | 71.1 [64.19 to 77.29]
  CS19F: number analyzed (Participants) | 198 | 201 | 200
  CS19F | 74.2 [67.59 to 80.18] | 72.1 [65.40 to 78.22] | 75.5 [68.94 to 81.29]
  CS22F: number analyzed (Participants) | 158 | 166 | 165
  CS22F | 76.6 [69.20 to 82.94] | 71.1 [63.55 to 77.85] | 14.5 [9.55 to 20.87]
  VS23F: number analyzed (Participants) | 194 | 185 | 190
  VS23F | 76.3 [69.67 to 82.09] | 81.1 [74.68 to 86.45] | 78.9 [72.46 to 84.51]
  VS33F: number analyzed (Participants) | 187 | 182 | 171
  VS33F | 53.5 [46.05 to 60.79] | 58.8 [51.27 to 66.02] | 8.8 [4.99 to 14.06]

9. Secondary Outcome: Percentage of Participants With a ≥4-fold Rise From Baseline in Geometric Mean Concentrations (GMCs) of Serotype-specific Immunoglobulin G (IgG) Antibodies
Description: The percentage of participants with ≥4-fold rise from baseline in IgG GMCs of each common serotype (CS) and V114-specific serotype (VS) were compared in the V114 and Prevnar® 13 arms. Estimated GMT, GMT ratio, 95% CI, and p-values were obtained from a constrained longitudinal data analysis (cLDA) model.
Time Frame: Baseline and Day 30 (one month after vaccination)
Population: All vaccinated participants with data available are included.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114-A | V114-B | Prevnar 13®
Number analyzed (Participants) | 231 | 231 | 227
Percentage of Participants
  CS1: number analyzed (Participants) | 216 | 215 | 214
  CS1 | 78.2 [72.14 to 83.55] | 69.8 [63.15 to 75.83] | 65.4 [58.63 to 71.77]
  CS3: number analyzed (Participants) | 216 | 215 | 214
  CS3 | 58.3 [51.45 to 64.98] | 46.5 [39.70 to 53.42] | 31.3 [25.16 to 37.98]
  CS4: number analyzed (Participants) | 216 | 215 | 214
  CS4 | 71.8 [65.25 to 77.66] | 63.7 [56.91 to 70.15] | 62.1 [55.29 to 68.67]
  CS5: number analyzed (Participants) | 216 | 215 | 214
  CS5 | 52.3 [45.43 to 59.13] | 47.0 [40.16 to 53.88] | 48.1 [41.27 to 55.04]
  CS6A: number analyzed (Participants) | 216 | 215 | 214
  CS6A | 73.6 [67.20 to 79.36] | 77.2 [71.01 to 82.64] | 77.1 [70.88 to 82.55]
  CS6B: number analyzed (Participants) | 216 | 215 | 214
  CS6B | 75.5 [69.17 to 81.05] | 77.2 [71.01 to 82.64] | 66.4 [59.60 to 72.65]
  CS7F: number analyzed (Participants) | 216 | 215 | 214
  CS7F | 69.4 [62.83 to 75.51] | 72.6 [66.08 to 78.41] | 69.6 [62.99 to 75.71]
  CS9V: number analyzed (Participants) | 216 | 215 | 214
  CS9V | 73.1 [64.77 to 77.23] | 71.6 [65.10 to 77.55] | 65.0 [58.15 to 71.33]
  CS14: number analyzed (Participants) | 216 | 215 | 214
  CS14 | 57.9 [50.98 to 64.54] | 48.8 [41.98 to 55.73] | 49.1 [42.19 to 55.97]
  CS18C: number analyzed (Participants) | 216 | 215 | 214
  CS18C | 71.8 [65.25 to 77.66] | 77.7 [71.51 to 83.06] | 70.6 [63.96 to 76.58]
  CS19A: number analyzed (Participants) | 216 | 215 | 214
  CS19A | 65.3 [58.52 to 71.61] | 67.9 [61.22 to 74.09] | 64.5 [57.67 to 70.89]
  CS19F: number analyzed (Participants) | 216 | 215 | 214
  CS19F | 59.7 [52.85 to 66.32] | 71.6 [65.10 to 77.55] | 62.6 [55.76 to 69.12]
  CS22F: number analyzed (Participants) | 216 | 215 | 214
  CS22F | 71.3 [64.77 to 77.23] | 71.2 [64.61 to 77.12] | 1.9 [0.51 to 4.72]
  VS23F: number analyzed (Participants) | 216 | 215 | 214
  VS23F | 72.2 [65.74 to 78.08] | 77.2 [71.01 to 82.64] | 71.5 [64.94 to 77.44]
  VS33F: number analyzed (Participants) | 216 | 215 | 214
  VS33F | 72.7 [66.23 to 78.51] | 65.6 [58.82 to 71.91] | 0.9 [0.11 to 3.34]

ADVERSE EVENTS:
Time Frame: Up to 30 days after vaccination
Description: All participants who received study vaccination are included.
Arm/Group | V114-A | V114-B | Prevnar 13®
All-Cause Mortality (participants affected / at risk) | 0/231 | 0/231 | 0/227
Serious Adverse Events (participants affected / at risk) | 1/231 | 2/231 | 0/227
Other Adverse Events (participants affected / at risk) | 169/231 | 163/231 | 148/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114-A (N=231) | V114-B (N=231) | Prevnar 13® (N=227)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114-A (N=231) | V114-B (N=231) | Prevnar 13® (N=227)
Fatigue (General disorders) | 56 (62) | 41 (44) | 51 (57)
Injection site erythema (General disorders) | 22 (22) | 29 (30) | 24 (24)
Injection site pain (General disorders) | 145 (159) | 140 (149) | 124 (134)
Injection site swelling (General disorders) | 29 (29) | 38 (38) | 29 (29)
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 (22) | 17 (17) | 14 (17)
Myalgia (Musculoskeletal and connective tissue disorders) | 53 (53) | 43 (45) | 32 (35)
Headache (Nervous system disorders) | 28 (34) | 29 (35) | 38 (41)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation.